CLINICAL TRIAL: NCT05166018
Title: Optimization of a Tool for Predicting Postoperative Clinical Evolution After Lumbar Surgery Multicenter Longitudinal Prospective Study on a National Cohort Clinical Evolution After Lumbar Surgery
Brief Title: Optimization of a Tool for Predicting Postoperative Clinical Evolution After Lumbar Surgery
Acronym: DeepSurgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cortexx Medical Intelligence (Industry)
Collaborators: Ramsay Générale de Santé (Other); Elsan (Other); Malakoff-Humanis (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DeepSurgeryMH_01
Record Dates: First submitted 2021-11-16; First posted 2021-12-21 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Spine Disease; Spinal Fusion; Surgery; Spine Degeneration
MeSH Terms: conditions — Spinal Diseases

STUDY DESIGN:
Intervention Model Description: The patient will be required to complete a guided digital questionnaire at each follow-up assessment.
  This questionnaire will be completed online by the patient in the Surgery Medical Outcomes (SuMO system) system developped by the Society Cortexx Medical Intelligence. The system access procedures and connection codes will be known to the patient by the investigating physician. Patients will, throughout the study, be automatically informed via the SUMO system of the availability of data to be completed. The security of patient data is guaranteed by encrypted and separate storage of medical data, in order to comply with applicable regulatory requirements.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SuMO Patient (Experimental): 92 data will be collected during the patient care episode. Among the 92 criteria, 63 are pre-operative, 29 are post-operative in order to provide an evolutionary prediction during the management of the patient.
  Post-operative follow-up criteria making it possible to establish the scalability or non-scalability of the quality of life after the surgical procedure.
  The results will be compared to the prediction proposed by the machine learning algorithm.
  Interventions: Diagnostic Test: SuMO Patient

INTERVENTIONS:
Diagnostic Test: SuMO Patient — The current study is interventional insofar as the patient is collecting all of his socio-medical information. The analysis of the data provided by the patient makes it possible to establish a long-term prognosis for the patient but does not in itself constitute a parallel medical approach.
  SUMO allows the surgeon to transmit post-operative advice developed by the surgeons themselves.

SUMMARY:
The objective of the study is the establishment, optimization and prospective evaluation of a digital predictive platform capable of providing for each lumbar spine operated patient a clinical predictive status: Patient green (success) orange (treatment failure ), red patient (complication) in order to optimize his medical care up to 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Major patient
* Eligible for lumbar decompression surgery, instrumented or not
* Social insured
* Having given consent
* Eligible for the acts described in Protocole

Exclusion Criteria:

* Minor
* Pregnant or breastfeeding woman
* Safeguard measure or guardianship
* Arthrodesis on more than 2 levels
* Interventions linked to a traumatic or infectious context are excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Optimization of a tool for predicting the postoperative clinical course after lumbar surgery | 14 months
  Establishment and prospective evaluation of a predictive tool with the area under the receiver operating characteristic (AUROC) metric >= 80% Sensitivity >= 90% Specificity >= 60% in the capacity of providing for each back operated patient a clinical predictive status: green patient (success) orange (treatment failure), red patient (complication).

SECONDARY OUTCOMES:
Collection of optimized data in the patient operative long terms care | 14 months
  Implementation, optimization and evaluation of a digital tool for collecting patient data on the episode of care
  Outcome (unit) - Result expected assessment time connection means preoperatively (second/connection) - 300s time 'use and navigation (second) - 1800s number of connections made by the patient preoperatively (number) - 5 number of connections / day before operation (number) - 1 number of use (number) - 15 number of drops / connection (Ratio%) - <20% number of lost view (no connection> 20 days) (Ratio%) - <10% evaluation of average using time post-operative (second/connections) - 300 Time of use and navigation (second) - 1800 number of connections made by the patient in post -operative (number) - 5 number of connections / day after operation (number)- 1 number of uses (number) - 15 number of withdrawals (Ratio%) - <20% number of lost to follow-up (no connection> 20 days) (Ratio%) - <10% number of documents analyzed / patient (number) - 10

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Polyclinique Jean Villar, Bruges, Nouvelle-Aquitaine
  - Clinique Geoffroy Saint-Hilaire, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Andre A, Peyrou B, Carpentier A, Vignaux JJ. Feasibility and Assessment of a Machine Learning-Based Predictive Model of Outcome After Lumbar Decompression Surgery. Global Spine J. 2022 Jun;12(5):894-908. doi: 10.1177/2192568220969373. Epub 2020 Nov 19. PMID 33207969
- See also: Mobile application for collecting patient's data — https://play.google.com/store/apps/details?id=com.sumoapp&hl=fr
- Available data/document: Individual Participant Data Set: SUMO — https://sumo.doc.cortexxmi.com/